CLINICAL TRIAL: NCT06637410
Title: Effectiveness of High Intensity Laser Treatment in Partial Supraspinatus Tendon Tears: A Randomised Controlled Trial
Brief Title: Effectiveness of High Intensity Laser Treatment In Partial Supraspinatus Tendon Tears
Acronym: HILT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Oznur Uzun, medical doctor, specialist of physical therapy and rehabilitation, deputy chief physician, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2-23-3841; Ankara Bilkent City Hospital (Other: Physical Medicine and Rehabilitation Hospital)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Shoulder Pain; Supraspinatus Tear
Keywords: HILT; rotator cuff; shoulder pain; supraspinatus; ultrasound
MeSH Terms: conditions — Shoulder Pain | interventions — Ultrasonic Therapy; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Group 1 (HILT group) received HILT 3 sessions per week for 3 weeks in addition to the therapeutic exercise program applied 5 sessions per week for 3 weeks. Group 2 (US group) received an ultrasound program 3 days a week in addition to a therapeutic exercise program of 5 sessions per week for 3 weeks. ROM exercises and Codman exercises, in a level not to increase the severity of the pain of the patient, were given and stretching and strengthening exercises were taught to the patients. They performed these exercises daily in two sets with five repeats in each set under the supervision of an experienced physiotherapist while taking their treatments.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HILT (HILT Group) (Experimental): HILT group received HILT 3 sessions per week for 3 weeks in addition to the therapeutic exercise program applied 5 sessions per week for 3 weeks. HILT was performed by a single physiotherapist experienced in using a laser device. In the HILT group, the device was used on the rotator cuff muscles in two stages: phase I and phase II. Pulse method was used in phase I for analgesic effect. For the biostimulation effect, the continuous wave method was used in phase II. In the next five sessions, biostimulation effect was applied using 7W power. A dose of 100 J/cm was applied longitudinally to the rotator cuff muscles area for a total energy of 2500 J for 25 minutes and 57 seconds up to 25 cm.
  Interventions: Device: High intensity laser therapy; Other: Therapeutic Exercise
- Ultrasound therapy (US Group) (Active Comparator): Ultrasound therapy was performed by a single physiotherapist experienced in using US device. US group received an ultrasound program 3 days a week in addition to a therapeutic exercise program of 5 sessions per week for 3 weeks. During US therapy, the patients were seated comfortably on chairs and their shoulders were in neutral position. The standard US dose was 1.2 W/cm2. The duration of ultrasound was 8 minutes. Using slow circular movements, the physiotherapist applied the transducer head of US device over the shoulder joint on an area of 25 cm2. US device was used in pulsed mode at a frequency of 1 MHz. The therapeutic ultrasound pulse cycle was 50%.
  Interventions: Device: Ultrasound therapy; Other: Therapeutic Exercise

INTERVENTIONS:
Device: High intensity laser therapy — HILT was performed by a single physiotherapist experienced in using a laser device. During HILT application, the patients were seated comfortably on chairs and their shoulders were in neutral position. The wavelength of the laser light used was 1064 nanometers. In the HILT group, the device was used on the rotator cuff muscles in two stages: phase I and phase II. Pulse method was used in phase I for analgesic effect. A standard frequency of 25 Hz is applied. During the first four therapy sessions, it was aimed to provide an analgesic effect by using 8 W power and 12 J/cm dose. The rays were applied to the rotator cuff muscles area in a circle from outside to inside for 2.5 minutes, for a total energy of 300 J, on an area of 25 cm2. For the biostimulation effect, the continuous wave method was used in phase II. n the next five sessions, biostimulation effect was applied using 7W power. A dose of 100 J/cm was applied longitudinally to the rotator cuff muscles.
  Arms: HILT (HILT Group)
Device: Ultrasound therapy — US therapy was performed by a single physiotherapist experienced in using US device. Calibration and control of the device are performed regularly. During US therapy, the patients were seated comfortably on chairs and their shoulders were in neutral position. The standard US dose was 1.2 W/cm2. The duration of ultrasound was 8 minutes. Using slow circular movements, the physiotherapist applied the transducer head of US device over the shoulder joint on an area of 25 cm2. US device was used in pulsed mode at a frequency of 1 MHz. The therapeutic ultrasound pulse cycle was 50%.
  Arms: Ultrasound therapy (US Group)
Other: Therapeutic Exercise — ROM exercises and Codman exercises, in a level not to increase the severity of the pain of the patient, were given and stretching and strengthening exercises were taught to the patients. They performed these exercises daily in two sets with five repeats in each set underCalibration and control of the device are performed regularly.

SUMMARY:
The primary goal of this clinical trial is to compare the effects of High Intensity Laser Therapy (HILT) on tears of tendons of shoulder girdle muscles with those of Ultrasound (US) therapy. It will also learn about the effects of HILT on pain and range of motion of injured shoulder. The main questions it aims to answer are:

Does HILT decrease the debilitating pain? Does HILT increase the range of motion of the sholuder joint? How long does the effect of HILT continue?

Researchers will compare the effects of HILT to a control group (ultrasound therapy group, an established method of treatment in shoulder girdle tendon tears) to see if HILT works better to treat shoulder girdle tendon tears.

Participants will:

receive HILT or US therapy 3 sessions per week for 3 weeks in addition to the therapeutic exercise program.

Visit the clinic at the beginning, at the 4th week and at the 12th week to determine the level of pain and disability via application of surveys.

Tendon thickness of participants will also be measured at the beginning, at the 4th week and at the 12th week to see if the treatment works to heal the tear.

DETAILED DESCRIPTION:
Shoulder disorders are one of the most common musculoskeletal problems worldwide. After low back pain and knee pain, shoulder pain has been estimated to be the third most common musculoskeletal presentation in primary care. Shoulder joint is surrounded by rotator cuff muscles and rotator cuff tendinopathy is the most common cause of shoulder pain. Shoulder pain caused by partial supraspinatus tendon tear (STT) is a complex and challenging issue for clinicians. The choice of the most appropriate treatment management for these tears is controversial.

For Ellman grade I and II tears which comprise STTs of less than 50% or tears which are below 6 mm in thickness, strengthening exercises, ultrasound (US) therapy, physical therapy, injection treatment and medical treatment can provide improvement in patients. However, in grade III tears which involve STTs of more than 50% of the muscle or tears above 6 mm in thickness surgical treatment may be required.

Recently, high-intensity laser therapy (HILT) has been introduced and used in treatment of musculoskeletal disorders. There is no universally accepted theory that explains the exact mechanism of the postulated laser effects, yet. Nd:YAG laser which has a wavelength of 1064 nm is used in HILT. It works in a therapeutic window that has a low absorbability rate in superficial tissue layers, so it penetrates more deeply than other types of lasers. In addition to having a higher power than low-intensity lasers, lasers used in HILT have a shorter laser emission time and a longer laser emission interval. Therefore, a large amount of laser irradiation can be delivered to deep tissues. The utilization of HILT has been expanding, and patients have reported significant improvement in function and reduction of pain.

To our knowledge, no studies to date have been conducted on the effects of HILT on partial STT. The aim of the present study was to evaluate the long-term effectiveness of HILT on pain, disability, and range of motion in patients with shoulder pain caused by STT and to compare its effects to those of US therapy.

The current study was designed as a prospective randomized controlled clinical trial and conducted after approval from the local ethics committee of our medical center. The study was conducted in accordance with the principles of Declaration of Helsinki and registered in the government database. The patients were recruited from the Ankara Bilkent City Hospital, physical medicine and rehabilitation outpatient clinic

ELIGIBILITY:
Inclusion Criteria:

* to be between 18-75 years old,
* the presence of shoulder pain for more than 3 months
* shoulder pain level of at least 3 on a 10-point Visual Analog Scale
* diagnosis of partial STT's which are below 6 mm in thickness
* no response to conservative treatments such as ice, soft tissue massage, stretching and nonsteroidal anti-inflammatory (NSAID) drugs after 6 weeks.

STT was detected with musculoskeletal system ultrasound by the same physician in outpatient clinic.

Exclusion Criteria:

* inflammatory rheumatic disease,
* cervical radiculopathy
* pregnancy,
* thyroid disease,
* history of cardiac pacemaker placement,
* epilepsy and/or any progressive neurological disease,
* history of shoulder surgery
* shoulder injection within the last 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) for pain | VAS for pain was applied to the patients before the procedure and at the 4th week and the 12th week after the procedure.
  VAS is used to measure musculoskeletal pain with very good reliability and validity (VAS, 0-10 cm; 0 means no pain, 10 means severe pain).

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | SPADI) was applied to the patients before the procedure and at the 4th week and 12th week after the procedure.
  Shoulder Pain and Disability Index (SPADI) was developed to measure shoulder discomfort. Its evaluation includes two parts: pain and disability. Part 1 includes five questions in the pain subgroup and measures the pain experienced by the patient over the previous week using VAS (0 no pain, to 10, most severe pain). Part 2 is the disability subgroup and includes eight questions and measures the degree of difficulty (0 no difficulty, to 10, requires help) in the movements of the patient during the last week.
  SPADI includes 13 questions, and zero point refers to maximal well-being and 130 points refers to maximal sickness. We evaluated each part of the SPADI; shoulder pain index (SPADI-SPI), shoulder disability index (SPADI-SDI) and total SPADI (SPADI-T) separately. Validity of SPADI was demonstrated in the literature. The Turkish version of the validity and reliability evaluation study for SPADI has already been implemented.
Supraspinatus tendon thickness | Supraspinatus tendon thickness was measured using ultrasonography before the study , four weeks after treatment , and 12 weeks later.
  Shoulder ultrasonography was performed on all patients using a 5-12 MHz linear array transducer by the same physician who was experienced in musculoskeletal system ultrasonography and was unaware of the patients' treatment group. Imaging was performed with the patient in a sitting position. The patient was asked to place the hand of the side under examination with the palm on the hip of the same side. (Modified Crass & Middleton position). While the arm was in extension and internal rotation positions, the probe was placed transversely to the lower part of the acromion, and the supraspinatus tendon and biceps tendon were seen in the same section. This image was frozen and 10-15-20 mm lateral from the end of the hyperechoic image of the biceps tendon was marked and supraspinatus tendon thickness was measured from these points.

CONTACTS AND LOCATIONS:
Overall Officials: Öznur Uzun, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Physical Medicine and Rehabilitation Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We can share our Study Protocol, Statistical Analysis plan and patients' informed Consent Forms.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD will become available starting 6 months after publication.
Access Criteria: The doctors who are specialized in Physical Medicine and Rehabilitation will be able to access upon contact with the principal investigators via email.

REFERENCES:
- [Result] Alayat MSM, Atya AM, Ali MME, Shousha TM. Correction to: Long-term effect of high-intensity laser therapy in the treatment of patients with chronic low back pain: a randomized blinded placebo-controlled trial. Lasers Med Sci. 2020 Feb;35(1):297. doi: 10.1007/s10103-019-02926-x. PMID 31788745
- [Result] Alayat MS, Mohamed AA, Helal OF, Khaled OA. Efficacy of high-intensity laser therapy in the treatment of chronic neck pain: a randomized double-blind placebo-control trial. Lasers Med Sci. 2016 May;31(4):687-94. doi: 10.1007/s10103-016-1910-2. Epub 2016 Feb 25. PMID 26914684
- [Result] Alayat MS, Elsodany AM, Miyajan AF, Alzhrani AA, Alzhrani HMS, Maqliyah AM. Changes in local skin temperature after the application of a pulsed Nd:YAG laser to healthy subjects: a prospective crossover controlled trial. Lasers Med Sci. 2019 Oct;34(8):1681-1688. doi: 10.1007/s10103-019-02769-6. Epub 2019 Mar 22. PMID 30903525
- [Result] Dundar U, Turkmen U, Toktas H, Solak O, Ulasli AM. Effect of high-intensity laser therapy in the management of myofascial pain syndrome of the trapezius: a double-blind, placebo-controlled study. Lasers Med Sci. 2015 Jan;30(1):325-32. doi: 10.1007/s10103-014-1671-8. Epub 2014 Oct 2. PMID 25274197
- [Result] Santamato A, Solfrizzi V, Panza F, Tondi G, Frisardi V, Leggin BG, Ranieri M, Fiore P. Short-term effects of high-intensity laser therapy versus ultrasound therapy in the treatment of people with subacromial impingement syndrome: a randomized clinical trial. Phys Ther. 2009 Jul;89(7):643-52. doi: 10.2522/ptj.20080139. Epub 2009 May 29. PMID 19482902
- [Result] Ellman H. Diagnosis and treatment of incomplete rotator cuff tears. Clin Orthop Relat Res. 1990 May;(254):64-74. PMID 2182260
- [Result] Mitchell C, Adebajo A, Hay E, Carr A. Shoulder pain: diagnosis and management in primary care. BMJ. 2005 Nov 12;331(7525):1124-8. doi: 10.1136/bmj.331.7525.1124. No abstract available. PMID 16282408
- [Result] Lucas J, van Doorn P, Hegedus E, Lewis J, van der Windt D. A systematic review of the global prevalence and incidence of shoulder pain. BMC Musculoskelet Disord. 2022 Dec 8;23(1):1073. doi: 10.1186/s12891-022-05973-8. PMID 36476476
- [Result] Castro BKC, Correa FG, Maia LB, Oliveira VC. Effectiveness of conservative therapy in tendinopathy-related shoulder pain: A systematic review of randomized controlled trials. Phys Ther Sport. 2021 May;49:15-20. doi: 10.1016/j.ptsp.2021.01.010. Epub 2021 Jan 28. PMID 33550201
- [Derived] Uzun O, Bilir EE, Arslan HB, Senturk B, Tezen O. Effectiveness of high intensity laser treatment in partial supraspinatus tendon tears: a randomised controlled trial. Lasers Med Sci. 2025 Jan 23;40(1):36. doi: 10.1007/s10103-025-04307-z. PMID 39849169